CLINICAL TRIAL: NCT07197580
Title: A Phase 3, Randomized, Multi-Center, Open-Label Study to Compare 177Lu-TLX250 (Lutetium (177Lu) Girentuximab Tetraxetan) With the Investigator's Choice of a Single Agent Therapy in Participants With Carbonic Anhydrase 9 (CAIX) Expressing, Advanced Relapsed or Recurrent Clear Cell Renal Cell Carcinoma (ccRCC)
Brief Title: Study of 177Lu-TLX250 in Advanced Relapsed or Recurrent ccRCC
Acronym: LUTEON
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Telix Pharmaceuticals (Innovations) Pty Limited (Industry)
Collaborators: Medpace, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 177Lu-TLX250-302
Record Dates: First submitted 2025-08-18; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: ccRCC; Renal Cell Carcinoma (Kidney Cancer); Renal Cell Carcinoma (RCC); Renal Cell Cancer Metastatic; Renal Cell Cancer, Recurrent; Clear Cell Renal Cell Cancer (ccRCC)
Keywords: Carbonic anhydrase 9; Clear Cell Renal Cell Cancer; Kidney Cancer; ccRCC; CA9; CA-9; CAIX; Girentuximab; CA9 target therapy; Positron-Emission Tomography; Radiation Therapy; Radiopharmaceuticals; Targeted Radiation
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 1887MBq 177Lu-girentuximab tetraxetan (Experimental): 3 infusions of 1887 MBq 177Lu-TLX250 at 8-week intervals or 6 infusions of 1258 MBq 177Lu-TLX250 at 4-week intervals (fractionation of 3 doses of 2516 MBq)
  Interventions: Radiation: 177Lu-TLX250
- 1258 MBq 177Lu-girentuximab tetraxetan (Experimental): 6 infusions of 1258 MBq 177Lu-TLX250 at 4-week intervals
  Interventions: Radiation: 177Lu-TLX250

INTERVENTIONS:
Radiation: 177Lu-TLX250 — 3 infusions of 177Lu-TLX250 at 8-week intervals or 6 infusions 177Lu-TLX250 at 4-week intervals
  Other Names: TLX250-Tx; 177Lu girentuximab tetraxetan

SUMMARY:
Multicenter Phase 3 study of 177Lu-TLX250 in adult participants with CAIX-expressing advanced, relapsed or recurrent clear cell renal cell carcinoma (ccRCC). Part 1 will evaluate two dosing regimens to determine the recommended Phase 3 dose (RP3D). Part 2 will compare 177Lu-TLX250 with investigator's choice of monotherapy aligned with Australian standard-of-care.

DETAILED DESCRIPTION:
This is a randomized, open-label, multi-center 3 study evaluating the safety and efficacy of 177Lu-TLX250, a CAIX-targeting radioligand therapy, in adult participants with advanced, relapsed or recurrent clear cell renal cell carcinoma (ccRCC).

The study consists of two parts:

• Part 1 (Phase 2a - Dose Optimization): Participants will be randomized to receive one of two dosing regimens of 177Lu-TLX250.

The objective of Part 1 is to determine the recommended Phase 3 dose (RP3D) for use in Part 2.

ELIGIBILITY:
Inclusion Criteria:

* be aged ≥ 18 years.
* have provided written informed consent, dated and signed by the participant prior to any study-specific procedure;
* have relapsed or recurrent, locally advanced, or metastatic RCC with histologically or cytologically confirmed diagnosis of RCC with clear cell component per American Joint Committee on Cancer Staging Manual (Edge SB et al., 2017), with or without sarcomatoid features;
* have received at least 2 and no more than 3 prior lines of systemic therapies for locally advanced or metastatic ccRCC including a PD-1/PD-L1 inhibitor (at least 2 administrations) and a VEGF/VEGFR-targeting agent (including TKI or mAb) in sequence or in combination;
* have had radiographic disease progression occurring during or after the most recent line of therapy or intolerance to most recent line of therapy;
* have at least one measurable lesion according to RECIST, version 1.1. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions;
* be CAIX-positive at Screening defined as having at least 1 lesion with a tumor-lesion CAIX ratio of the maximum standardized uptake value (SUVmax) to liver mean standardized uptake value SUVmean) ≥ 1.5 as determined by BICR of 89Zr-TLX250 PET outcomes;
* have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 to 1;
* have recovered from the AEs related to prior lines of therapy or returned to baseline with the exception of Grade 2 neurotoxicity. Ongoing, controlled AEs, such as hypothyroidism or hypertension, are permitted;
* have adequate organ function, defined as:
* Bone Marrow:

  * leukocytes ≥ 3,000/µL;
  * absolute neutrophil count ≥ 1500/µL (administration of granulocyte colony stimulating factor is not allowed within 4 weeks prior to the first administration of 177Lu-TLX250;
  * platelets ≥ 100,000/µL (platelet transfusion is not allowed within 4 weeks prior to the first administration of 177Lu-TLX250); and
  * hemoglobin ≥ 9g/dL (red blood cell transfusion is not allowed within 2 weeks prior to the first administration of 177Lu-TLX250).
* Liver Function:

  * total bilirubin ≤ 1.5 × the upper limit of normal (ULN). For patients with known Gilbert's Syndrome ≤ 3 × ULN is permitted; and
  * alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN or ≤ 5.0 × ULN for participants with liver metastases.
* Renal Function:

  * creatinine clearance ≥ 40 mL/min as measured by Cockroft-Gault formula or directly calculated by 24h urine;
  * have negative pregnancy test for women of childbearing potential (serum); and

Exclusion Criteria:

* have any of the following:

  * visceral metastatic lesions that are ≥ 1 cm that have a CAIX TLR < 1;
  * lytic bone metastatic lesions with a soft tissue component of at least 1 cm with a TLR < 1; and/or
  * at least one metastatic lymph node lesion with short axis ≥ 2.5 cm with a TLR <1;
* received prior 177Lu-TLX250 therapy, any other radioligand therapy, or any prior CAIX-targeting therapy;
* have any known hypersensitivity to compounds of similar chemical or biologic composition to girentuximab, DFO or DOTA linker, zirconium or lutetium, and/or any excipient in the study drug or radiographic contrast-agents;
* has received G-CSF or erythropoietin within 4 weeks prior to laboratory evaluations at Screening;
* be currently receiving or have received:

  * any radionuclide within 10 half-lives of the radionuclide prior to 89Zr-TLX250 administration;
  * any type of systemic anticancer therapy within 2 weeks before the first administration of 177Lu-TLX250;
  * prior radiotherapy within 2 weeks prior to the first administration of 177Lu-TLX250 (must have recovered from all radiation-related toxicities and not currently require steroid treatment); and/or
  * prior palliative radiation (≤2 weeks of radiotherapy) within 1-week of the first administration of 177Lu-TLX250 for non-central nervous system disease; NOTE: If the investigator feels that the patient is continuing to receive some clinical benefit from standard-of-care (SOC) therapy, the patient may continue SOC therapy up until 2 weeks prior to dosing with 177Lu-TLX250.
* have known brain metastases, unless these have been treated and stabilized for at least 4 weeks prior to the first administration of 177Lu-TLX250; Note: Participants with a history of brain metastases must have either a head CT with contrast-or brain MRI performed at Screening to document stable disease prior to the first administration of 177LuTLX250.
* Have experienced any major trauma including major surgery (such as abdominal/ cardiac/thoracic surgery) within 3 weeks of administration of the first administration of 177LuTLX250;
* be pregnant or intend to become pregnant, breastfeed, or conceive a child during the study period and for at least 42 days after last administration of 89Zr-TLX250 or 6 months after last administration of 177Lu-TLX250, depending on which study drug is administered last to the respective participant;
* Note: Contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies (see Appendix 10.4).
* be planning to breastfeed during the study period and for 28 days after last administration of 89ZrTLX250 or 75 days after last administration of 177Lu-TLX250, depending on which study drug is administered last to the respective participant;
* have active and uncontrolled infections requiring systemic therapy or other severe concurrent disease, which, in the opinion of the investigator, would place the participant at undue risk or interfere with the study;
* have a history of concurrent malignancy with a life expectancy of ≤ 2 years or requirement of systemic anti-cancer therapy or requirement of local therapy that would confound study results; however; participants with the following malignancies can be enrolled into the study:

  * basal cell or squamous cell carcinoma of the skin;
  * carcinoma in situ of the cervix, breast or bladder; and/or
  * incidental histologic finding of prostate cancer;
* have a serious, non-healing wound, ulcer, or bone fracture;
* be unable to stay in the scanner bed with the arms resting out of the thoracic and abdominal fields (i.e., arms alongside the body or raised arm position) for the duration of the scan;
* have not had resolution of clinically significant toxic effects of prior systemic cancer therapy, surgery, or radiotherapy to Grade ≤1 (except for laboratory parameters specified above, Grade 2 alopecia, and/or stable Grade 2 sensory neuropathy, according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0;
* have inflammatory bowel disease (e.g. Crohn's disease, ulcerative colitis, etc.);
* have a life expectancy shorter than 3 months;
* have bleeding or thrombotic disorders or subjects at risk for severe hemorrhage;
* have experienced any clinically significant bleeding, including hemoptysis or tumor bleeding within 2 weeks prior to the first administration of 177Lu-TLX250;
* has evidence of a serious active or sub-clinical infection or angina pectoris (New York Heart Association [NYHA] Class III or IV), significantly prolonged QT interval or other serious illness(es) involving the cardiac, respiratory, central nervous system, renal, hepatic or hematological organ systems, that might impair the ability to complete this study or could interfere with determination of causality of any adverse effects experienced in this study, or which require treatment that could interact with study treatment; or
* have any medical or other condition that in the opinion of the investigator(s) would preclude the subject's participation in a clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Dose Optimization -safety and tolerability | Through study completion, an average of 1.5 years
  Part 1 of the study is being done to identify the best dose to use for Part 2 of the study.
  Assessing adverse events of special interest (AESIs), incidence and severity of treatment-emergent adverse events (TEAEs) and frequency, severity according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) V5.0, seriousness, and relationship of study treatment will be assessed. Laboratory abnormalities will be assessed according to the NCI CTCAE V5.0.
Efficacy- median mPFS | Through study completion, an average of 2 years
  Primary objective for Part 2 of the study and secondary objective for Part 1. Monitoring disease progression according to Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1).

SECONDARY OUTCOMES:
Monitoring OS (Overall Survival) | Through study completion, an average of 2 years
  Time from the date of randomization to death from any cause
Monitoring ORR (Objective Response Rate) | Through study completion, an average of 2 years
  Proportion of participants achieving confirmed objective response rate (ORR), i.e., complete response (CR) or partial response (PR) per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) as assessed by a blinded independent central review (BICR)
Monitoring DoR (Duration of Response) | Through study completion, an average of 2 years
  Time from the first documentation of objective response, i.e., complete response (CR) or partial response (PR) to the first documentation of disease progression or death due to any cause as assessed by blinded independent central review (BICR)
Monitoring DCR (Disease control Rate) | Through study completion, an average of 2 years
  The proportion of participants achieving confirmed objective response, i.e., complete response (CR), partial response (PR), or stable disease (SD) per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) as assessed by blinded independent central review (BICR)
Evaluate blood radioactive PK parameter- Cmax (maximum plasma concentration) | Treatment period (4 months)
  Gamma-counting blood radioactivity will be used to derive this pharmacokinetics parameter
Evaluate blood radioactive PK parameter- AUCinf (area under blood concentration time curve from zero to infinity) | During Treatment (4 months)
  Gamma-counting blood radioactivity will be used to derive this pharmacokinetics parameter.
Evaluate blood radioactive PK parameter- t1/2 (Terminal half-life) | During Treatment (4 months)
  Gamma-counting blood radioactivity will be used to derive this pharmacokinetics parameter.
Evaluate blood radioactive PK parameter- CL (Clearance) | During Treatment (4 months)
  Gamma-counting blood radioactivity will be used to derive this pharmacokinetics parameter.
Tumor and Organ-specific 177Lu-TLX250 absorbed radiation values | During Treatment (4 months)
  Images-radiation values for tumor and lesions will be measured and analyzed after first and second administration of 177Lu-TLX250.
TAC for tumor and organ | During Treatment (4 months)
  Time Activity Curves (TAC) will be used to derive time integrated activity parameters in tumor and organ
Tumor- and organ-specific 177Lu-TLX250 residence time | During Treatment (4 months)
  Residence time of 177Lu-TLX250 in tumor and organs will be derived and interpreted
Identification of dose-limiting organ(s) | During Treatment (4 months)
  Absorbed dose will be compared to maximal dosimetry threshold for each organ to evaluated the dose limiting organ
Characterize health utility as measured using the European Quality of Life 5 Dimensions 5 Level Version (EuroQoL EQ-5D-5L) | Through study completion, an average of 2 years
  Health utility scores from the European Quality of Life 5 Dimensions 5 Level Version (EuroQoL EQ-5D-5L) questionnaire
Change from Baseline in EORTC QLQ-C30 Physical Functioning | Through study completion, an average of 2 years
  Assessed using the EORTC QLQ-C30 questionnaire to evaluate physical functioning.
Change from Baseline in EORTC QLQ-C30 Global Health Status/HRQoL | Through study completion, an average of 2 years
  Assessed using the EORTC QLQ-C30 questionnaire to evaluate overall health-related quality of life.
Change from Baseline in FKSI-DRS Subscale | Through study completion, an average of 2 years
  Assessed using the FKSI-DRS (Functional Assessment of Cancer Therapy - Kidney Symptom Index) to evaluate disease-related symptoms.
Incidence and Severity of AESIs and TEAEs | Through study completion, an average of 2 years
  Adverse events will be assessed and graded per NCI-CTCAE v5.0 criteria.
Dosing Delays Due to 177Lu-TLX250-Related TEAEs | Through study completion, an average of 2 years
  Number of dosing delays attributed to TEAEs related to 177Lu-TLX250.
Activity Level Reductions Due to 177Lu-TLX250-Related TEAEs | Through study completion, an average of 2 years
  Number of participants with reduced activity levels due to TEAEs related to 177Lu-TLX250.
Evaluation of Immunogenicity (HACA) | Through study completion, an average of 2 years
  Incidence of HACA positivity, overall per treatment group, and per visit (to track incidence over time)
Evaluation of HACA on PK/Biodistribution | Through study completion, an average of 2 years
  Evaluate any correlation of incidence of HACA positivity to changes in PK/Biodistribution per treatment group
Evaluation of HACA on efficacy/safety | Through study completion, an average of 2 years
  Evaluate any correlation of incidence of HACA positivity to changes in efficacy/safety end points per treatment group
Characterization of HACA neutralizing activity | Through study completion, an average of 2 years
  For confirmed positive HACA samples, incidence of nAb positivity, overall per treatment group, and per visit (to track incidence over time), as applicable
Evaluation of nAb on PK/Biodistribution | Through study completion, an average of 2 years
  Evaluate any correlation of incidence of nAb positivity to changes in PK/Biodistribution per treatment group
Evaluation of nAB on efficacy/safety | Through study completion, an average of 2 years
  Evaluate any correlation of incidence of nAb positivity to changes in efficacy/safety end points per treatment group
Evaluate Radiation Exposure-Response parameter- normalized absorbed dose to individual organs (mGy/MBq) | Through study completion, an average of 2 years
  Evaluate relationship between normalized absorbed dose to individual organs with DCR, ORR and incidence and severity of AESI
Evaluate Radiation Exposure-Response parameter- AUC | Through study completion, an average of 2 years
  Evaluate relationship between AUC to individual organs with DCR, ORR and incidence and severity of AESI.
Evaluate Radiation Exposure-Response parameter- Cmax | Through study completion, an average of 2 years
  Evaluate relationship between Cmax to individual organs with DCR, ORR and incidence and severity of AESI.
Evaluate Radiation Exposure-Response parameter- normalized absorbed dose to tumors (mGy/MBq) | Through study completion, an average of 2 years
  Evaluate relationship between normalized absorbed dose to tumor with DCR, ORR and incidence and severity of AESI.

CONTACTS AND LOCATIONS:
Locations (3):
- Australia (3):
  - Austin Health, Heidelberg, Victoria
  - Melbourne Theranostic Innovation Centre (MTIC), Melbourne N., Victoria
  - GenesisCare, Fiona Stanley Hospital (Murdoch), Murdoch, Washington

IPD SHARING:
Plan to Share IPD: No
We have opted not to share individual participant data due to concerns regarding participant privacy and the absence of explicit consent for data sharing in the original trial protocol.

REFERENCES:
- [Result] Muselaers CH, Boers-Sonderen MJ, van Oostenbrugge TJ, Boerman OC, Desar IM, Stillebroer AB, Mulder SF, van Herpen CM, Langenhuijsen JF, Oosterwijk E, Oyen WJ, Mulders PF. Phase 2 Study of Lutetium 177-Labeled Anti-Carbonic Anhydrase IX Monoclonal Antibody Girentuximab in Patients with Advanced Renal Cell Carcinoma. Eur Urol. 2016 May;69(5):767-70. doi: 10.1016/j.eururo.2015.11.033. Epub 2015 Dec 23. PMID 26706103
- [Result] Stillebroer AB, Boerman OC, Desar IM, Boers-Sonderen MJ, van Herpen CM, Langenhuijsen JF, Smith-Jones PM, Oosterwijk E, Oyen WJ, Mulders PF. Phase 1 radioimmunotherapy study with lutetium 177-labeled anti-carbonic anhydrase IX monoclonal antibody girentuximab in patients with advanced renal cell carcinoma. Eur Urol. 2013 Sep;64(3):478-85. doi: 10.1016/j.eururo.2012.08.024. Epub 2012 Aug 21. PMID 22980441